CLINICAL TRIAL: NCT04963127
Title: Prospective Observational Study of Diagnostic Accuracy of Dual-Energy-/Multi-Energy-CT for the Detection of Bone Marrow Edema
Brief Title: Prospective Study of Diagnostic Accuracy of Spectral CT for the Detection of Bone Marrow Edema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0318
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Fractures, Bone; Bone Marrow Edema
Keywords: Spectral CT; Multi-Energy CT; Dual-Energy CT; Bone Marrow Edema
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: 400 patients who are scheduled to undergo a clinically requested CT scan of parts of the skeleton using a Dual-Energy/Multi-Energy/Spectral acquisition mode to exclude or further define bone fractures.
  Interventions: Diagnostic Test: Computed Tomography of the skeleton using a Dual-Energy-/Multi-Energy-/Spectral acquisition mode
- Retrospective Cohort: 400 patients who had undergone a clinically requested CT scan of the skeleton in standard acquisition mode in the past to exclude or further define bone fractures.
  Interventions: Diagnostic Test: Computed Tomography of the skeleton using a conventional single-energy / non-spectral acquisition mode

INTERVENTIONS:
Diagnostic Test: Computed Tomography of the skeleton using a Dual-Energy-/Multi-Energy-/Spectral acquisition mode — CT acquisition using a Dual-Energy / Multi-Energy / Spectral acquisition mode
  Other Names: Spectral Imaging
  Groups: Prospective Cohort
Diagnostic Test: Computed Tomography of the skeleton using a conventional single-energy / non-spectral acquisition mode — CT acquisition using a standard single energy / non-spectral acquisition mode
  Groups: Retrospective Cohort

SUMMARY:
Dual-Energy/Multi-Energy/Spectral-CT can visualize bone marrow edema associated with fractures, however, current scientific evidence is mostly derived from to retrospective analyses. Our prospective study systematically analyzes the diagnostic accuracy of the visualization of bone marrow edema by including patients who are scheduled for a CT scan to exclude or further characterize a fracture. After giving informed consent, the CT scan will be performed using a dose-neutral Dual-Energy-/Multi-Energy-/Spectral-CT acquisition technique. If the patient undergoes MRI of the same region within 7 days, this scan will be used as a gold-standard for bone marrow edema. This will allow the quantification of diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion for a fracture AND
* indication for CT confirmed by board-certified radiologist ('justified indication' according to German/European radiation protection law) AND
* patient (is able to give informed consent and) has given informed consent.

Exclusion Criteria:

* cardiorespiratory instability (as judged by the referring physician)
* age < 18 years
* known or suspected pregnancy
* known bone metastases of a malignant disease
* known rheumatic disease
* metal implants in the region to be scanned
* surgical intervention over the last 12 months in the region to be scanned
* contraindications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at least 18 years of age who are referred by the emergency department for a CT scan with the suspicion of a fracture.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Dual-Energy/Multi-Energy/Spectral CT to detect bone marrow edema in comparison with MRI as the goldstandard. | MRI of the same region can be used for comparison if performed within 7 days
  sensitivity, specificity and positive and negative likelihood ratios will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Schwarz, MD, Principal Investigator — University Hospital Augsburg
Locations (1):
- University Hospital Augsburg, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data upon request (pending final approval by the data protection officer of the university hospital).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Requests for sharing individual participant data will be considered at the time of publication of the first manuscript containing result data.
Access Criteria: We plan to share data on request at this point in time.